CLINICAL TRIAL: NCT04284852
Title: Niraparib Maintenance in Patients With Advanced Ovarian Cancer at Neoadjuvant Setting - a Phase 2, Single-arm Trial (NEOPRIMA Trial)
Brief Title: Niraparib Maintenance in Patients With Advanced Ovarian Cancer at Neoadjuvant Setting
Acronym: NEOPRIMA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW-19-681
Record Dates: First submitted 2020-02-17; First posted 2020-02-26 (Actual); Last update posted 2023-12-15 (Actual); Status verified 2023-10

CONDITIONS: Ovarian Cancer
Keywords: advanced; ovarian; cancer; neoadjuvant; niraparib
MeSH Terms: conditions — Ovarian Neoplasms; Neoplasms | interventions — niraparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Niraparib 200 or 300mg daily orally for 18 cycles unless disease progression or intolerable side effects (whichever occurs first)
  Interventions: Drug: Niraparib

INTERVENTIONS:
Drug: Niraparib — PARP inhibitor
  Other Names: Zejula

SUMMARY:
This study aims to evaluate the effects of niraparib in those who have received neoadjuvant chemotherapy and subsequent interval debulking surgery, with or without hyperthermic intraperitoneal chemotherapy, and would also explore if there are any biomarkers, other than BRCA / HRD status and platinum sensitivity, that may help to identify those who may benefit from PARPi especially those who are HRD negative.

DETAILED DESCRIPTION:
Despite cytoreductive surgery and platinum-based chemotherapy, about 70% of patients with advanced ovarian cancer recur in the first 2 - 3 years. PARPi has been shown to be prolong survival in primary advanced ovarian cancer. However its role in neoadjuvant setting has not been fully evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be at least 18 years old.
2. Patients must have newly diagnosed, histologically confirmed high grade, serous or endometrioid, FIGO stage 3 or 4, ovarian, fallopian tube or primary peritoneal carcinoma before the start of NACT.
3. Patients must have received 3 - 4 cycles of NACT containing either carboplatin or cisplatin, IDS with or without HIPEC, and 3 - 6 more cycles of adjuvant chemotherapy, prior to recruitment into the study.
4. The patients should have only one cytoreductive surgery.
5. The patients must show either complete (CR) or partial response (PR) to the platinum-based chemotherapy using RECIST 1.1 criteria.
6. Patients should not be amenable to further surgery or radiotherapy except for the purpose of symptomatic relief.
7. All surgery, chemotherapy and radiotherapy should finish more than 3 weeks prior to recruitment.
8. Niraparib should be started within 8 weeks after the last dose of chemotherapy.
9. Patients should have Eastern Cooperative Oncology Group (ECOG) performance score 0 to 2 within 28 days prior to recruitment.
10. Patients must have adequate bone marrow, renal, hepatic and neurological function within 28 days prior to the start of treatment.
11. Patients who have childbearing potential should practice highly effective contraception throughout the study until at least 30 days after completion of the treatment.

Exclusion Criteria:

1. Patients who are diagnosed to have low-grade or borderline carcinoma, mucinous or clear cell cystadenocarcinoma, carcinosarcoma or undifferentiated carcinoma, are excluded.
2. Patients who have stable disease or PD on the post-treatment scan or clinical evidence are excluded.
3. Patients who have drainage of ascites within 4 weeks before recruitment are excluded.
4. Patients who have with concurrent malignancy within five years (except for basal or squamous cell skin cancer or in-situ breast cancer) are excluded.
5. Patients who have history of unresolved thrombocytopenia, myelodysplastic syndrome or acute myeloid leukaemia are excluded.
6. Patients who have symptomatic brain or leptomeningeal metastases, or spinal cord compression are excluded unless these are treated and controlled within 28 days of recruitment.
7. Patients with the significant past medical history, such as active hepatitis, myocardiac infarction, in the last six months are excluded.
8. Patients with severe gastrointestinal conditions such as evidence of bowel obstruction in the last 4 weeks prior to enrolment, or history of inflammatory bowel disease, are not eligible.
9. Patients having had severe infections within 4 weeks prior to the start of treatment are excluded.
10. Patents with active tuberculosis, history of positive test for human immunodeficiency virus (HIV) or known acquired immunodeficiency syndrome (AIDS) are excluded.
11. Patients with prior allogeneic stem cell or solid organ transplantation are excluded.
12. Those patients who suffer from CTCAE grade 2 or more toxicity from previous treatment, except alopecia, are excluded.
13. Patients who have used PARPi previously are excluded.
14. Patients who are allergic to any component of niraparib are excluded.
15. Patients who have used bevacizumab, or who are going to use bevacizumab as maintenance, are not eligible to join the study.
16. Use of other investigational drugs within 28 days or at least 5 half-lives (whichever is longer) before study drug administration is not allowed.
17. Patients who are pregnant or breastfeeding are excluded.
18. Patients must not have either platelet or red blood cell transfusion, or granulocyte colony stimulating factor (G-CSF) within 2 weeks of the first dose of study treatment.
19. Patients must not plan to donate blood during the study or for 90 days after the last dose of study treatment.
20. Patients with major operation within 28 days or open biopsy within 7 days before enrolment are not eligible.
21. Patients planned to have major surgery during the course of the study are excluded.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Actual)
Dates: Start 2020-05-01 (Actual); Primary Completion 2023-10-01 (Actual); Study Completion 2023-10-01 (Actual)

PRIMARY OUTCOMES:
PFS rate at 18 months | up to 18 months
  Proportion of patients who are progression-free at 18 months according to the RECIST 1.1

SECONDARY OUTCOMES:
PFS by the RECIST 1.1 | up to 5 years
  The time from first dose of trial medication to first documentation of objective tumor progression (PD) or to death due to any cause, whichever occurs first.
Overall survival | up to 5 years
  Overall survival is defined as the time from first dose of trial medication to date of death due to any cause.
OS rate at 18 months | up to 18 months
  Proportion of patients who are alive at 18 months
Change of biomarkers | up to 18 months
  Expression levels of markers like Ki-67 before and after chemotherapy
Treatment-related adverse events | up to 18 months
  Incidence of treatment-related adverse events classified by CTCAE version 5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ka Yu Tse, FRCOG, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No